CLINICAL TRIAL: NCT01238289
Title: Peer-Led Diabetes Education Programs in High Risk Mexican Americans Evaluates Glycemic Control Compared to Standard Approaches: A Project Dulce™ Promotora Randomized Trial
Brief Title: Randomized Trial of Peer Led Education-Project Dulce
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH); San Diego State University (Other)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Corp VP, Scripps Whittier Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R18DK070666-01A1 (NIH); R18DK070666-01A1 (NIH)
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Type 2 Diabetes
Keywords: peer education; diabetes; randomized; trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): This arm continues with standard care at community clinic
  Interventions: Behavioral: Control
- Peer Education (Experimental): This group receives 8 weeks of peer led self management education classes and subsequent monthly support groups for a total of 10 months
  Interventions: Behavioral: Peer Education

INTERVENTIONS:
Behavioral: Peer Education — Conduct peer education classes for 8 weeks and support groups monthly for a total of 10 months and evaluate effects on metabolic and behavior outcomes
  Other Names: Project Dulce
  Arms: Peer Education
Behavioral: Control — This group continues with standard care at the community health center
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the effect of a culturally sensitive diabetes self-management program on glucose control and metabolic parameters in low income Mexican-Americans with type 2 diabetes using the Project Dulce model utilizing a low cost, peer-educator format.

DETAILED DESCRIPTION:
To recruit 207 Mexican-Americans patients from federally-funded community health centers in San Diego County with Hemoglobin A1c (HbA1c) > 8% and randomize to Project Dulce peer intervention or continuation of standard diabetes care. The primary outcome will be the percent change in HbA1c levels at 10 months following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Mexican American, men and women, 21-75 years old, who were under-insured patients at federally qualified community health centers in San Diego County with type 2 diabetes and HbA1c > or = 8%.

Exclusion Criteria:

* Individuals with a physical or mental health condition that would preclude fulfilling the requirements of the study were ineligible to participate, HbA1c < 8,pregnant with gestational diabetes

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2006-09; Primary Completion 2009-03 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
mean percent change Hemoglobin A1c (HbA1c) | Baseline, 4 months and 10 months
  Evaluate change in HbA1c over a 10 month time period from baseline.

SECONDARY OUTCOMES:
Body mass index, blood pressure and lipid changes | Baseline, 4 months and 10 months
  Evaluate change in Body mass index, blood pressure and lipids over a 10 month time period from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Whittier Diabetes Institute
Locations (1):
- Scripps Whittier Diabetes Institute, La Jolla, California, United States